CLINICAL TRIAL: NCT06653647
Title: Pilot Efficacy of a Guided Imagery Therapy Mobile Application for Functional Abdominal Pain Disorders in Children
Brief Title: Efficacy of Guided Imagery Therapy Mobile Application for Functional Abdominal Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John M Hollier, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-51406; K23DK120928 (NIH)
Record Dates: First submitted 2024-09-17; First posted 2024-10-22 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Functional Abdominal Pain Disorders; Irritable Bowel Syndrome (IBS); Functional Gastrointestinal Disorders; Functional Colonic Disease; Gastrointestinal Disease; Digestive System Diseases; Neurological Manifestations; Signs and Symptoms, Digestive; Pain; Abdominal Pain/ Discomfort
Keywords: abdominal pain; irritable bowel syndrome; recurrent abdominal pain
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases; Colonic Diseases, Functional; Digestive System Diseases; Neurologic Manifestations; Signs and Symptoms, Digestive; Pain; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: Qualified participants will be randomized into either the Delayed Treatment group or the Immediate Treatment Group. The Delayed Treatment Group will be observed for the first 8 weeks after randomization, and then outcome data will be reassessed through abdominal pain and stool diaries and other surveys. Then, this group will be crossed over to the treatment phase and given access to the mobile app intervention for another eight weeks. After this 8-week intervention phase, outcomes will be reassessed again via an abdominal pain and stooling diary and other surveys.
  Those qualified participants randomized to the Immediate Treatment Group will be given access to the mobile app intervention for eight weeks. At the end of the eight weeks, outcome measures will be reassessed through an abdominal pain and stooling diary and other surveys.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Active Comparator): Participants randomized to the Immediate Treatment arm will receive immediate access to the guided imagery therapy mobile application intervention.
  Interventions: Behavioral: Guided Imagery Therapy
- Delayed Treatment (Other): Participants randomized to the Delayed Treatment arm will be placed on waitlist status and will not have any intervention from weeks 3 to 10. Participants will continue their usual care for their abdominal pain during this time. Then, this study arm will cross over to the guided imagery therapy mobile application intervention from weeks 11 to 18.
  Interventions: Behavioral: Guided Imagery Therapy

INTERVENTIONS:
Behavioral: Guided Imagery Therapy — Participants will be asked to listen to a pre-recorded, 10 to 15 minute guided imagery therapy (GIT) session via mobile application 5 out of 7 days per week for 8 weeks in addition to their usual care for their abdominal pain.

SUMMARY:
Chronic abdominal pain is common among children, and the majority of cases are attributed to functional abdominal pain disorders. One approach to treating these disorders is by using psychological therapies. This clinical trial aims to see how well pre-recorded guided imagery therapy sessions help children's abdominal pain when delivered via a mobile application (app) on a smartphone or tablet.

Participants will complete a baseline abdominal pain and stooling diary to determine eligibility and other surveys. Participants who qualify will be placed in one of two groups by chance:

* Immediate Treatment Group
* Delayed Treatment Group

After randomization, the Immediate Treatment Group will get immediate access to the guided imagery therapy (GIT) mobile app intervention. This intervention asks participants to listen to a 10- to 15-minute GIT session 5 out 7 days weekly for 8 weeks in addition to their usual care for their abdominal pain. Then, participants will complete another abdominal pain and stooling diary and other psychometric surveys at the end of this intervention period.

After randomization, the Delayed Treatment group will be observed as they wait 8 weeks without app access. During this phase, these participants will continue to treat their abdominal pain in their usual fashion. After the end of this waiting period, participants will complete another abdominal pain and stooling diary and psychometric surveys again before gaining access to the GIT mobile app intervention. As noted previously, the mobile app intervention will ask participants to listen to a 10- to 15-minute GIT session 5 out of 7 days weekly for 8 weeks in addition to their usual care for their abdominal pain. Another abdominal pain and stooling diary and other psychometric surveys will be collected at the end of this app intervention.

DETAILED DESCRIPTION:
After fully disclosing the study design, intervention options, randomization scheme, and potential side effects of the interventions, caregivers and their children will document their respective informed consent and assent electronically. REDCap is a secure web application designed for surveys and databases. All data captured through REDCap will be encrypted and transmitted securely to HIPAA-compliant institutional servers for storage.

Participants and their caregivers will complete the following surveys at baseline, second baseline phase (delayed treatment group only 8 weeks after baseline), and immediately post-therapy (delayed treatment group 16 weeks after baseline and immediate treatment group 8 weeks after baseline) through REDCap:

* 2-week Abdominal Pain and Stooling Diary
* Children's Somatic Symptoms Inventory (child self-report and parent proxy-report)
* Pain Catastrophizing Scale - Child Version
* Pain Catastrophizing Scale - Parent Version
* Pediatric Quality of Life Inventory 4.0 Generic Core (child self-report and parent proxy-report)
* Behavior Assessment System for Children 3rd Ed (child self-report and parent proxy-report)

ELIGIBILITY:
Study staff will enroll children with functional abdominal pain disorders and their primary caregiver for this study.

Inclusion Criteria:

* Texas Children's Pediatrics patients 7 to 12 years old at enrollment
* A Rome IV Functional Abdominal Pain Disorder as defined by a 2-week abdominal pain and stooling diary
* Both children and their primary caregivers must be able to read and communicate in English proficiently to understand the intervention's audio therapy sessions and psychometric instruments.

Exclusion Criteria:

* Prior participation in principal investigator's related feasibility or usability study
* Previous abdominal surgeries
* Co-morbid conditions associated with abdominal pain (e.g., cystic fibrosis)
* Autism
* Significant development delay
* Psychosis
* Prior experience with cognitive behavioral therapy or guided imagery therapy to treat chronic abdominal pain
* Alarm symptoms that warrant further medical evaluation (e.g., blood in stool)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2025-07-18 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain Frequency | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Average number of abdominal pain episodes per day from a self-report 2-week abdominal pain diary

SECONDARY OUTCOMES:
Abdominal Pain Intensity | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Average daily abdominal pain severity measured on a 0-10 (10 is most severe) ordinal scale from a self-report 2-week abdominal pain diary
Anxiety | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Behavior Assessment System for Children, third edition, child self-report Anxiety Scale, t score ranges from 20 to 120, higher scores are worse
Anxiety | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Behavior Assessment System for Children, third edition, parent proxy-report Anxiety Scale, t score ranges from 20 to 120, higher scores are worse
Depression | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Behavior Assessment System for Children, third edition, child self-report Depression scale, t score ranges from 20 to 120, higher scores are worse
Depression | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Behavior Assessment System for Children, third edition, parent-proxy report Depression scale, t scores ranges from 20 to 120, higher scores are worse
Somatization | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Children's Somatic Symptoms Inventory child self-report, raw score ranges from 0 to 96, higher scores are worse
Somatization | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Children's Somatic Symptoms Inventory parent-proxy report, raw score ranges from 0 to 96, higher scores are worse
Pain Catastrophizing Thoughts | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Pain Catastrophizing Scale - Child Version, raw score ranges from 0 to 52, higher scores are worse
Pain Catastrophizing Thoughts | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Pain Catastrophizing Scale - Parent Version, raw score range from 0 to 52, higher scores are worse
Health-Related Quality of Life | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Pediatric Quality of Life Inventory Generic Core Scales 4.0 child self-report, raw score ranges from 0 to 100, higher scores are better
Health-Related Quality of Life | Baseline (both groups), Second baseline (delayed treatment group only, 8 weeks after baseline), and Post-intervention (delayed group 16 weeks after initial baseline, immediate group 8 weeks after baseline)
  Pediatric Quality of Life Inventory Generic Core Scales 4.0 parent-proxy report, raw score ranges from 0 to 100, higher scores are better

CONTACTS AND LOCATIONS:
Overall Officials: John M Hollier, MD, MS, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine / Texas Children's Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No